CLINICAL TRIAL: NCT00543582
Title: A Phase 2, Open-label Trial to Evaluate the Efficacy and Safety of MGCD0103 Administered in Combination With Azacitidine (Vidaza®) to Subjects With Relapsed or Refractory Hodgkin or Non-Hodgkin Lymphoma, and to Evaluate the Pharmacokinetics of Different Formulations of MGCD0103
Brief Title: MGCD0103 Administered in Combination With Azacitidine (Vidaza®) to Subjects With Relapsed or Refractory Hodgkin or Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Celgene terminated its collaboration agreement with MethylGene for the development of MGCD0103. All Celgene-sponsored trials with MGCD0103 will be closed.
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103 PH US 2007 CL002
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Hodgkin Lymphoma; Non-Hodgkin Lymphoma (Follicular or Large Diffuse B-cell Lymphoma or Mantle Cell Lymphoma)
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell | interventions — mocetinostat; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MGCD0103 and Azacitidine

INTERVENTIONS:
Drug: MGCD0103 and Azacitidine — In Part 1 of the study, up to 22 people to enroll will receive a single, oral dose (75 mg gelcap) of MGCD0103 and FB-MGCD0103 during their first 2 weeks in the study. Up to 22 additional people will receive a single dose of both MGCD0103 and TA-FB-MGCE0103. The next group of people to enroll will receive 2 different single doses (25, 50, 100 mg) of FB-MGCD0103 or TA-FB-MGCD0103 during their first 2 weeks in the study.
  In Part 2 of the study, from Day 1-5 of each 28-day cycle, all subjects will receive a dose of azacitidine (75 mg/m2) either subcutaneously or through an intravenous device, and on days 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, a single, oral dose (85 mg) of MGCD0103 until progression or unacceptable toxicity develops.
  Other Names: Vidaza®

SUMMARY:
The first part of the study is to evaluate and determine if three different forms of MGCD0103 (free base FB-MGCD0103, tartaric acid free base [TA-FB-MGCD0103], and dihydrobromide [2HBr] salt formulation MGCD0103) have the same properties when given to patients with cancer. The second part of the study is to determine whether MGCD0103 administered in combination with azacitidine is effective and safe in treating subjects with relapsed or refractory Hodgkin's lymphoma or non-Hodgkin's lymphoma (NHL) (follicular or diffuse large B-cell [DLBCL]).

DETAILED DESCRIPTION:
MGCD0103 and FB-MGCD0103 belong to a class of drugs known as histone deacetylase inhibitors (also called HDAC inhibitors). Azacitidine belongs to a class of anti-cancer drugs known as DNA de-methylating agents. Azacitidine (Vidaza®) was approved by the Food and Drug Administration (FDA) in 2004 for the treatment of myelodysplastic syndromes (MDS).

The combination of MGCD0103 and azacitidine has been given to about 50 people with leukemia or MDS in other clinical studies. This is the first study where the combination will be tested in people with lymphoma. Specifically, the study is designed to understand the following:

* How long single doses of TA-FB-MGCD0103, FB-MGCD0103 and MGCD0103 stay in the body, OR
* How long different doses of TA-FB-MGCD0103 and FB-MGCD0103 stay in the body; and
* How long MGCD0103 stays in the body when given with azacitidine; and
* What effect MGCD0103 and azacitidine have on the body and the study subject's type of lymphoma; and
* If the genetic and chemical make-up of the study subject's blood and/or tumor play a role in how she/he responds or does not respond to MGCD0103 and azacitidine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically confirmed diagnosis of classical Hodgkin's lymphoma or NHL (follicular, DLBCL, or mantle cell) and confirmed relapsed or refractory disease. 1)Subjects with a diagnosis of classical Hodgkin's lymphoma MUST have relapsed following a prior autologous, allogeneic or reduced intensity allogeneic stem cell transplant. Subjects who received an allogeneic transplant must have no evidence of graft versus host disease (GVHD), and have discontinued treatment with immunosuppressive agents ≥ 3 months prior to enrollment in this study. 2)Subjects with DLBCL must be ineligible for, or have refused, autologous stem cell transplant, or have relapsed following transplant. 3)Subjects with MCL must have relapsed after prior treatment and not be eligible for autologous stem cell transplant (ASCT) or have relapsed following ASCT. 4)Subjects with NHL who may have received a prior allogeneic stem cell transplant must have no evidence of GVHD, and have discontinued treatment with immunosuppressive agents ≥ 3 months prior to enrollment in this study.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2 Evidence of measurable disease (ie, at least one lesion that can accurately be measured in at least two dimensions as ≥15 mm with spiral CT scan). 1)If only single target lesion must be PET positive, and measure ≥20mm in two dimensions (required only for subjects with Hodgkin's lymphoma and DLBCL).
* Adequate organ function including: 1)Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (≥1500/mm^3); and 2)Platelets ≥ 50 x 10^9/L (≥50,000/mm^3); and 3)Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (unless increased due to Gilbert's Syndrome or hemolysis); and 4)AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN; and 5)Serum creatinine ≤ 1.5 x ULN.
* At least 3 weeks elapsed since any prior anticancer therapy (standard or investigational) and full recovery (NCI CTCAE grade 1) from the toxic effects of that treatment.
* For women of childbearing potential, a negative serum pregnancy test within 7 days of treatment, a negative urine pregnancy test immediately prior to the first treatment with study drugs, and use of 2 physician-approved methods of birth control throughout the study and for a period of 3 months following the study.
* Written informed consent, willingness, and ability to comply with all study procedures.

Exclusion Criteria:

* Prior HDAC inhibitor and azacitidine combination therapy.
* Known hypersensitivity to azacitidine, HDAC inhibitors, and/or any components of MGCD0103, FB-MGCD0103, or TA-FB-MGCD0103 capsules and or azacitidine formulation components.
* Any condition that will put the subject at undue risk or discomfort as a result of adherence to study procedures (eg, requirement to take MGCD0103 with Gatorade®).
* Previous or concurrent malignancy except adequately treated basal cell or squamous skin cancer; in situ carcinoma of the cervix, or other solid tumor treated curatively, and without evidence of recurrence for at least 3 years prior to study entry.
* Presence of significant involvement of the liver by lymphoma and impaired synthetic function as indicated by hypoalbuminemia of < 1.0 x LLN.
* Active and uncontrolled clinically significant infection.
* Known Hepatitis B surface antigen (HepB SAg) positive or Hepatitis C antibody positive.
* Known infection with human immunodeficiency virus (HIV).
* History of melena or hematemesis within the last 3 months.
* Known central nervous system metastases.
* Less than 4 weeks elapsed since any major surgery.
* Pregnant or lactating women. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of beginning Part 1 of the study.
* WOCBP and men whose partners are WOCBP must use two acceptable methods of contraception while enrolled in this study, and for a period of 3 months following study drug treatment. Subjects unwilling or unable to follow this guideline will be excluded.
* Concurrent chronic treatment with therapeutic doses of systemic steroids.
* Prior or active disease or conditions that, in the opinion of the investigator, may interfere with the procedures or evaluations to be conducted in the study. This includes, but is not limited to, uncontrolled intercurrent illnesses such as symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Primary efficacy is measured by: 1) PET, CT & physical exam, 2) overall response rate (complete response=disease is gone, partial response=disease has improved). Study treatment continues as long as the cancer is stable & side effects are tolerable. | every other cycle of 28 days each

SECONDARY OUTCOMES:
Duration of response defined as: 1)the time of first documented objective response (either complete response or partial response) until the subject's disease gets worse, 2)how long his/her disease is stable. | 28 days after the last study drug

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reid, MSc, MBA, Study Director — MethylGene Inc.
Locations (4):
- United States (4):
  - St. Francis Cancer Research Foundation, Beech Grove, Indiana
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Weill Medical College of Cornell University, New York, New York
  - University of Texas, MD Anderson, Houston, Texas